CLINICAL TRIAL: NCT00001072
Title: A Phase I Safety and Immunogenicity Trial of Live Recombinant Canarypox ALVAC-HIV vCP300 and HIV-1 SF-2 rgp120 in HIV-1 Uninfected Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Prevention
Other Study IDs: AVEG 026; 10576 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Vaccines, Synthetic; HIV Envelope Protein gp120; AIDS Vaccines; HIV Seronegativity; Avipoxvirus; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Biological: ALVAC-HIV MN120TMGNP (vCP300)
Biological: ALVAC-RG Rabies Glycoprotein (vCP65)
Biological: rgp120/HIV-1 SF-2

SUMMARY:
To evaluate, in HIV-negative volunteers, the safety and immunogenicity of ALVAC-HIV MN120TMGNP (vCP300) followed by or combined with boosting using rgp120/HIV-1SF2. To compare ALVAC-HIV vCP300 with ALVAC-RG rabies glycoprotein (vCP65) as a control. To evaluate an accelerated immunization schedule at 0, 1, 3, and 6 months versus 0, 1, 6, and 9 months.

The combination of a live recombinant primer followed by a subunit boost has the potential to induce not only cytotoxic T lymphocytes but also neutralizing antibody.

DETAILED DESCRIPTION:
The combination of a live recombinant primer followed by a subunit boost has the potential to induce not only cytotoxic T lymphocytes but also neutralizing antibody.

Volunteers are randomized to one of seven groups to receive immunizations with either ALVAC-HIV vCP300 or ALVAC-RG vCP65 (control), plus simultaneous or sequential boosting with rgp120/HIV-1SF2 or placebo. Immunizations are given at 0, 1, 6, and 9 months or 0, 1, 3, and 6 months. Volunteers are followed for at least 24 months.

ELIGIBILITY:
Inclusion Criteria

Volunteers must have:

* Normal history and physical exam.
* ELISA and Western blot negative for HIV.
* CD4 count >= 400 cells/mm3.
* Normal urine dipstick with esterase and nitrite.
* Lower risk sexual behavior.

Exclusion Criteria

Co-existing Condition:

Subjects with the following symptoms or conditions are excluded:

* Positive hepatitis B surface antigen.
* Medical or psychiatric condition (such as recent suicidal ideation or present psychosis) that precludes compliance.
* Active syphilis. NOTE: Subjects with serology documented to be a false positive or due to a remote (> 6 months) treated infection are eligible.
* Active tuberculosis. NOTE: Subjects with a positive PPD and a normal chest x-ray showing no evidence of TB and not requiring isoniazid therapy are eligible.
* Allergy to egg products or neomycin.

Subjects with the following prior conditions are excluded:

* History of immunodeficiency, chronic illness, autoimmune disease, or use of immunosuppressive medications.
* History of anaphylaxis or other serious adverse reactions to vaccines.
* Prior immunization against rabies.
* History of serious allergic reaction to any substance, requiring hospitalization or emergent medical care (e.g., Stevens-Johnson syndrome, bronchospasm, or hypotension).
* Prior psychiatric condition (such as history of suicide attempts or past psychosis) that precludes compliance.
* History of cancer unless there has been surgical excision that is considered to have achieved cure.

Prior Medication:

Excluded:

* Live attenuated vaccines within 60 days prior to study entry. NOTE: Medically indicated killed or subunit vaccines (e.g., influenza, pneumococcal) do not exclude if administered at least 2 weeks from HIV immunizations.
* Experimental agents within 30 days prior to study entry.
* Prior HIV vaccines.
* Prior rabies immunization.

Prior Treatment:

Excluded:

* Blood products or immunoglobulin within 6 months prior to study entry. Identifiable high-risk behavior for HIV infection, such as
* injection drug use within past 12 months.
* higher or intermediate risk sexual behavior.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140
Dates: Study Completion 1999-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keefer M, Study Chair; Evans T, Study Chair
Locations (6):
- United States (6):
  - UAB AVEG, Birmingham, Alabama
  - JHU AVEG, Baltimore, Maryland
  - St. Louis Univ. School of Medicine AVEG, St Louis, Missouri
  - Univ. of Rochester AVEG, Rochester, New York
  - Vanderbilt Univ. Hosp. AVEG, Nashville, Tennessee
  - UW - Seattle AVEG, Seattle, Washington

REFERENCES:
- [Background] Evans TG, Keefer MC, Wolff M, Weinhold K, Excler JL, Duliege AM, McNamara J, McElrath JM, Graham BJ, Clements ML, Mulligan M, Belshe RB, Tartaglia J. Immunization of HIV-1 non-infected volunteers with a canarypox recombinant containing HIV-1 env, gag, pol, and nef genes (vCP 300) given simultaneously or followed by recombinant HIV-1 SF2 gp120. Conf Retroviruses Opportunistic Infect. 1997 Jan 22-26;4th:204 (abstract no 754)
- [Background] Gorse GJ, Patel GB, Mandava MD, Belshe RB. Vaccine-induced cytotoxic T lymphocytes against human immunodeficiency virus type 1 using two complementary in vitro stimulation strategies. Vaccine. 1999 Dec 10;18(9-10):835-49. doi: 10.1016/s0264-410x(99)00323-0. PMID 10580197
- [Background] Evans T, Corey L, Clements-Mann ML, Weinhold K, Belshe RB, Excler JL, Duliege AM. CD8+ CTL induced in AIDS vaccine evaluation group phase I trials using canarypox vectors (ALVAC) encoding multiple HIV gene products (vCP125, vCP205, vCP300) given with or without subunit boost. Int Conf AIDS. 1998;12:277 (abstract no 495/21192)
- [Background] Castillo RC, Arango-Jaramllo S, Humphrey W, Weinhold K, Schwartz DH. Vaccine induced CTL activity correlates with resistant phenotype in an in vitro challenge system. Conf Retroviruses Opportunistic Infect. 1998 Feb 1-5;5th:95 (abstract no 91)
- [Background] Evans TG, Keefer MC, Weinhold KJ, Wolff M, Montefiori D, Gorse GJ, Graham BS, McElrath MJ, Clements-Mann ML, Mulligan MJ, Fast P, Walker MC, Excler JL, Duliege AM, Tartaglia J. A canarypox vaccine expressing multiple human immunodeficiency virus type 1 genes given alone or with rgp120 elicits broad and durable CD8+ cytotoxic T lymphocyte responses in seronegative volunteers. J Infect Dis. 1999 Aug;180(2):290-8. doi: 10.1086/314895. PMID 10395842
- [Background] Sabbaj S, Corey L, Evans T, Keefer M, Excler JL, Duliege AM, Mulligan MJ, McGhee JR. Cytokine profiles in human PBMC T cell cultures stimulated with HIV antigens in seronegative volunteers immunized with canarypox expressing HIV antigens and boosted with recombinant SF2 GP120. Conf Adv AIDS Vaccine Dev. 1997 May 4-7:215 (Poster 110)
- [Background] Kaslow RA, Rivers C, Goepfert P, Tang J, El Habib R, Weinhold K, Mulligan MJ. Association of HLA class I alleles with cytotoxic T-lymphocyte (CTL) responses to gag and env in recipients of ALVAC-HIV canarypox vaccines. 7th Conference on Retroviruses and Opportunistic Infections. 2000 Jan 30-Feb 2 [Poster 818]
- [Background] Bender TJ, Tang J, Rivers C, Mulligan MJ, Kaslow RA. Grouping by HLA class I supertype does not enhance HLA associations with CTL responses to ALVAC-HIV canarypox vaccine components. 8th Conf Retro and Opportun Infect. 2001 Feb 4-8 (abstract no 193)